CLINICAL TRIAL: NCT00123084
Title: Efficacy of Voice Treatment for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DC001150 (NIH); R01DC001150 (NIH)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2017-04

CONDITIONS: Parkinson's Disease; Dysphagia; Dysarthria
Keywords: Parkinson's disease; Swallowing difficulties; speech; voice
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders; Dysarthria; Speech | interventions — Voice

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Voice/Respiratory Treatment (Experimental): 4 Days a week for 4 weeks with focus on high intensity voice exercises
  Interventions: Behavioral: Voice/Respiration Treatment
- Articulation Treatment (Experimental): 4 days a week for 4 weeks with focus on high intensity articulation tasks
  Interventions: Behavioral: Speech/Articulation Treatment
- Subjects with PD in a no treatment group (No Intervention): Subjects do not receive therapy during experimental phases, and will be offered therapy at the end of the study enrollment period.
- Healthy Control Subjects (No Intervention): Subjects are without Parkinson disease and will not receive therapy.

INTERVENTIONS:
Behavioral: Voice/Respiration Treatment — Therapy is 4 1-hour sessions per week for 4 weeks. Tasks include high-effort exercises focusing on increased loudness and good voice quality.
  Other Names: LSVT LOUD
  Arms: Voice/Respiratory Treatment
Behavioral: Speech/Articulation Treatment — Therapy is 4 1-hour sessions per week for 4 weeks. Tasks include high-effort articulation exercises to promote more enunciated speech.
  Other Names: LSVT ARTIC
  Arms: Articulation Treatment

SUMMARY:
The purpose of the research study is to determine the effects of two different kinds of speech treatment on certain behaviors in individuals with parkinson's disease. These behaviors include speech, voice, related communication behaviors, swallowing and body movement.

DETAILED DESCRIPTION:
This is a research project designed to look at various areas of function, such as speech, voice, swallowing, related communication behaviors and body movement of individuals with idiopathic Parkinson disease (PD) and to investigate how two different forms of speech therapy affect these areas.

We are asking up to 620 individuals to participate in this study in several different ways. Specifically, there is an experimental group (ExpG), questionnaire group (QG) and communication partner group (CPG). The ExpG will be composed of individuals with PD and the healthy age and gender matched controls (HC)(Up to 140 total will be asked, 80 expected to complete the study). The QG will include the significant others, family members, and friends of the ExpG (Up to 140 will be asked, 80 expected to complete the study). The CPG will be made up of friends of the ExpG (Up to 340 will be asked, 240 expected to complete the study).Some individuals in the ExpG may not pass the initial screenings. As a result, their QG and CPG will no longer need to participate. Therefore, the actual number of individuals who will complete the study is expected to be much less.

There are 10 PHASES of this study. The initial PHASES (1,2,3) are screening PHASES to determine if the individual is a good candidate for this study. PHASES 4, 6 and 10 are PHASES of recording data and PHASE 5 is treatment. PHASES 7, 8 and 9 are additional assessments. The total duration of the Subjects (Ss) participation from the time Ss sign the consent to the completion of the last phase (PHASE 10) is approximately10 months.

PHASE 1: ENT/CLINICAL VOICE AND SPEECH SCREEN PHASE 2: SWALLOW SCREEN AND ASSESSMENT PHASE 3: THINKING SKILLS SCREEN AND ASSESSMENT After the completion of PHASES 1-3, the research team will look at the data collected and determine if the Ss meet the criteria to participate in this study. If asked to participate, Ss will be assigned to one of four groups and then continue with PHASE 4.

PHASE 4: INITIAL DATA RECORDINGS All of the procedures in PHASE 4 will be done two times before the treatment PHASE 5. Each recording will take approximately 2-2.5 hours.

PHASE 5: TREATMENT PHASE 6: POST TREATMENT PHASE DATA RECORDINGS PHASE 7: FOLLOW-UP ENT EVALUATION PHASE 8: FOLLOW-UP SWALLOW EVALUATION PHASE 9: FOLLOW-UP THINKING SKILLS EVALUATION PHASE 10: 6-MONTH POST TREATMENT PHASE DATA RECORDINGS

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease (IPD)
* None or mild dementia
* None, mild or moderate depression
* Mild, moderate or severe speech, voice, and swallowing disorder

Exclusion Criteria:

* Severe depression
* Moderate or severe dementia
* Symptoms of another neurological condition other than or in addition to IPD or drug abuse
* Head or neck cancer
* Significant history of gastrointestinal disease or surgery
* Speech or voice disorders unrelated to IPD
* Neurosurgery, not for management of PD symptoms
* Laryngeal pathology/surgery
* Full-course Lee Silverman Voice Treatment (LSVT®)
* Smoked in last four years
* Absence of speech, voice or swallowing disorder
* Severe temporomandibular joint disorder
* Pregnancy (or the possibility of pregnancy)
* Hearing loss unexpected for his/her chronological age

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2002-03; Primary Completion 2012-09-30 (Actual); Study Completion 2012-09-30 (Actual)

PRIMARY OUTCOMES:
Voice intensity; voice fundamental frequency; articulatory acoustics; physiological voice function; speech intelligibility; swallowing function; non-verbal communication behaviors; limb function; neural imaging; neuropsychological functioning | 8-9 months

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Ramig, PhD, CCC-SLP, Principal Investigator — Professor, University of Colorado-Boulder; Senior Scientist, National Center for Voice and Speech-Denver; Adjunct Professor, Columbia University-NYC
Locations (2):
- United States (2):
  - National Center for Voice and Speech-Denver; An Affiliate of the unniversity of Colorado, Denver, Colorado
  - University of Texas HSC San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Levy ES, Moya-Gale G, Chang YHM, Freeman K, Forrest K, Brin MF, Ramig LA. The effects of intensive speech treatment on intelligibility in Parkinson's disease: A randomised controlled trial. EClinicalMedicine. 2020 Jun 28;24:100429. doi: 10.1016/j.eclinm.2020.100429. eCollection 2020 Jul. PMID 32639484